CLINICAL TRIAL: NCT01965236
Title: Influence of Sodium Intake on Left Ventricular-arterial Coupling in Hypertension: Biomechanical Assessment and Modelisation of Left Ventricular Function With Arterial Pressure
Brief Title: Influence of Sodium Intake on Left Ventricular-arterial Coupling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8985
Record Dates: First submitted 2013-10-08; First posted 2013-10-18 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
Keywords: hypertension, sodium intake, left ventricular function
MeSH Terms: conditions — Hypertension | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Patients are given 5 pills (1 g per pill) of sodium chloride per day for 6 weeks. After a one-week wash out period, a second period of 6 weeks is started with 5 placebo (microcrystalline cellulose) pills per day.
  Interventions: Dietary Supplement: sodium chloride; Dietary Supplement: Placebo
- Group 2 (Experimental): Patients are given 5 placebo (microcrystalline cellulose) pills per day for 6 weeks. After a one-week wash out period, a second period of 6 weeks is started with 5 pills (1 g per pill) of sodium chloride per day.
  Interventions: Dietary Supplement: sodium chloride; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: sodium chloride — Patients are given 5 pills (1 g per pill) of sodium chloride per day for 6 weeks. After a one-week wash out period, a second period of 6 weeks is started with 5 placebo (microcrystalline cellulose) pills per day.
Dietary Supplement: Placebo

SUMMARY:
The objective of the present study is to asses the effectiveness of the aorta-ventricular coupling according to low and high sodium intake in 28 controled hypertensive patients.

DETAILED DESCRIPTION:
Comparison of left ventricular function in two groups of 13 patients according to their different salt's consumption in double blind and crossover study. Performance estimation of the left ventricle by echocardiographic and central arterial pressure by tonometry.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension stage 1, with medium or high risk, when the treatment (mono or therapy without diuretics) is efficient, when the great pressure is reached (<140/90 mmHg)
* High sodium intake (sodium urinary excretion for 24h (UNaV) > or = 170 mmol/24h before visit 0
* Limited sodium intake objective (UNaV<85 mmol/24h)attempted at the end of the limited sodium intake period of 2 weeks
* Patients aged between 18 and 80 years
* Subject has given written informed consent
* Subject has subscribed a health care insurance

Exclusion Criteria:

* Secondary hypertension
* Complications associated with the arterial hypertension : history of cardiovascular diseases or myocardial infarction, cerebrovascular accident, coronary disease, ...
* Arterial hypertension associated with cardiopathy
* Arterial hypertension associated with nephropathy
* Arterial hypertension associated with diabetes
* Measure of central arterial pressure by tonometry is impossible
* Cardiac echogenicity is not satisfactory for the analysis of left ventricular loop analysis
* Patient refuses informed consent
* Follow-up impossible for 15 weeks
* Pregnant or women without efficacy contraception
* Patient without freedom by administration decision
* Patient in exclusion period
* Patient without french insurance
* Adult protected by the law

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
ultrasound volume, imaging "strain" and tonometry | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem DU CAYLAR, Principal Investigator — Department of intern Medicine and arterial Hypertension Lapeyronie University Hospital of Montpellier, Montpellier, France, 34295
Locations (1):
- Lapeyronie University Hospital of Montpellier, Montpellier, France